CLINICAL TRIAL: NCT00529074
Title: Epidural Anesthesia /Analgesia Versus PCA for Laparoscopic Complex Ventral Hernia Repair: A Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never activated
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO-1053537
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-05

CONDITIONS: Analgesia
Keywords: Epidural Analgesia
MeSH Terms: conditions — Agnosia | interventions — Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Epidural Catheter for Analgesia — Patients enrolled will be placed into one of two groups of 30 patients. The decision to place the patients in either one of the two groups will be randomized as above. The Epidural group will have a thoracic epidural catheter placed pre-operatively at the T6-T7 level before general anesthesia is given. (using a .1% Marcaine and .1% Meperidine solution) A dose of Ketorolac will be given 15 minutes before the patient will be awakened from anesthesia (provided that there is good renal function and the patient is not hypovolemic) The catheter will be used preoperatively as an adjunct for general anesthesia as well as used postoperatively for continuous epidural analgesia(CEA). The control group will be given general anesthesia alone and post-operative PCA along with NSAIDS before leaving for the recovery room (as above).

SUMMARY:
We plan to demonstrate the superiority of epidural anaesthesia/analgesia in repairs of large ventral hernias as compared with a conventional narcotic analgesia regimen.

We hypothesize that:

1. Primary outcome measures will improve. Patients will have a shorter length of stay (1 day less) with pre and post-operative epidural analgesia.
2. Secondary outcome measures will also improve. Among them will be VAS pain scores, time to first flatus and bowel movement as well as major and minor complications.

DETAILED DESCRIPTION:
Epidural anesthesia and analgesia has shown benefits over standard anesthesia/analgesia in many types of Vascular, GI, and Thoracic surgeries. The benefits extended are varied, and include: improvements in cardiac and pulmonary function, decreases in hypercoagulability, reduction of post-operative ileus and decreases in post-operative pain. 1 Epidural pain relief works by exposing the epidural space, with its network of nerve roots, to a flood of analgesics and/or local anesthetic. This is thought to prevent the release of neurotransmitters from afferent pain fibers or interrupt the transmission of pain related information to the dorsal horn of the spinal cord. 2 Several studies have been done on patients undergoing GI surgery with adjunct epidurals (particularly colorectal procedures) and they have shown that ileus and length of stay, is greatly reduced. 3No one has yet extended these benefits to patients undergoing hernia repair.

Laparoscopic ventral hernia repair has recently become a popular choice for both patients and surgeons alike, and has been shown in some studies to reduce wound complications and length of hospital stay. But improvements in post-operative pain, ileus and return to work have been less than hoped for, and as such, adjuncts are being investigated to improve some of these outcomes. In one study of 850 patients in 4 different academic institutions patients had a mean hospital stay of 2.3 days (although a great portion of cases were small ventral hernias that resulted in same-day discharges) and 3% remained hospitalized with a prolonged ileus. The proportion of patients who had prolonged ileus and subsequently longer hospital stays was much greater amongst the patients with larger ventral hernia repairs as well as the patients with recurrences.4 Moreover there has been some suggestion by Ramshaw and colleagues that Laparoscopic Ventral hernia repair is more painful than the classical open hernia operation. 5 One of the explanations is that there may be a component of parietal as well as visceral pain to this procedure; with the visceral pain accompanying the counter-traction on the herniated contents of the sac when taking down adhesions, and the parietal pain from the many full thickness sutures and 3mm tacks used to secure the prosthesis into the abdominal wall.6 In this study, we will test the benefits of epidural anesthesia/analgesia on these patients with complicated Laparoscopic ventral hernia repairs.

As of yet there have been no studies that compare the use of epidural analgesia/anesthesia to conventional anesthesia and narcotics for these patients in relation to their expected length of stay, post-op pain, ileus, or other complications.

1. Moraca RJ, Sheldon DG, Thirlby RC The role of Epidural Anesthesia and Analgesia in Surgical Practice. Annals of Surgery 2003;238 663-673.
2. R. J. Fotiadis1, S. Badvie1, M. D.Weston2 and T. G. Allen-Mersh1 Epidural analgesia in gastrointestinal surgery British Journal of Surgery 2004; 91: 828-841
3. Rodgers A, Walker N et al. Reduction of Post Operative Mortality and Morbidity With Epidural or Spinal Anaesthesia: Results From an Overview of Randomized Trials. Br Med Journal 2000; 321: 1493-1497
4. Heniford BT. Park A. Ramshaw BJ. Voeller G. Laparoscopic repair of ventral hernias: nine years' experience with 850 consecutive hernias. Annals of Surgery. 238(3):391-9; discussion 399-400, 2003 Sep
5. Ramshaw B, Esartia Et Al.Comparison of Laparoscopic and open Ventral Hernia Repair; The American Surgeon; Sept 1999; Vol 65: 9 pg 827
6. Heniford BT, Park, A, ramshaw BJ, Voeller G Laparoscopic Ventral Hernia Repair in 407 Patients. Journal of the American College of Surgeons. Vol 190: 6 PP 645-650 June 2000

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* ASA grades I-III
* Patients with large hernias

  1. requiring mesh greater than or equal to 18cmx 30cm
  2. with a known hernia of at least 10cm x 8cm
  3. Or several smaller hernias that require or may require the coverage referred to in #1

Exclusion Criteria:

* Age<18 or >80
* Poor candidacy for operative treatment
* Previous spinal operations
* Sepsis
* Incarcerated ventral hernias requiring anticoagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures will improve. Patients will have a shorter length of stay (1 day less) with pre and post-operative epidural analgesia. | Post-operatively

SECONDARY OUTCOMES:
Secondary outcome measures will also improve. Among them will be VAS pain scores, time to first flatus and bowel movement as well as major and minor complications. | Post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ramshaw, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States